CLINICAL TRIAL: NCT00023361
Title: TBTC Study 23: Treatment of HIV-Related Tuberculosis Using a Rifabutin-Based Regimen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDC-NCHSTP-2174; TBTC STUDY 23
Record Dates: First submitted 2001-09-06; First posted 2001-09-10 (Estimated); Last update posted 2005-09-05 (Estimated); Status verified 2005-09

CONDITIONS: HIV Infections; Tuberculosis
Keywords: tuberculosis; TB
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — Rifabutin

INTERVENTIONS:
Drug: Rifabutin

SUMMARY:
Primary objective:

To determine the rate of confirmed treatment failure and relapse with an intermittent rifabutin-based regimen for the treatment of isoniazid and rifamycin-susceptible HIV-related tuberculosis (TB).

ELIGIBILITY:
Inclusion Criteria

* Clinical diagnosis of pulmonary &/or extrapulmonary TB confirmed by a positive culture and susceptibility to rifampin. Patients having isoniazid or pyrazinamide (PZA)-resistant isolates are eligible to continue in the study on a modified regimen
* Evidence of HIV infection confirmed by a positive serologic test (ELISA and Western Blot).
* Absolute neutrophil count >500/mm3 (use of colony stimulating factors, filgrastim, or sargramostim is allowed)
* > 18 years of age
* Willingness to practice effective contraception if applicable
* Signed informed consent

Exclusion Criteria

* Pregnancy or breastfeeding
* AST > 10 times the upper limit of normal
* Bilirubin > 3.0 times the upper limit of normal
* Creatinine > 3.0 times the upper limit of normal
* Intolerance to any of the study drugs except isoniazid or pyrazinamide
* Concomitant disorder that is contraindication to the use of the study drugs
* More than 28 days of treatment for active tuberculosis within the 6 months prior to this course of therapy
* Bone/joint tuberculosis or silicotuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215
Dates: Start 1999-02; Study Completion 2003-02

PRIMARY OUTCOMES:
Rate of confirmed treatment failure and relapse

SECONDARY OUTCOMES:
Safety and tolerability
Response of HIV RNA to TB treatment
Paradoxical reactions

CONTACTS AND LOCATIONS:
Overall Officials: William Burman, MD, Study Chair — Denver Health and Hospitals
Locations (23):
- United States (20):
  - Central Arkansas Veterans Health System, Little Rock, Arkansas
  - LA County/USC Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Denver Department of Public Health and Hospitals, Denver, Colorado
  - Washington, D.C. VAMC, Washington D.C., District of Columbia
  - Chicago VA Medical Center (Lakeside), Chicago, Illinois
  - Hines VA Medical Center, Hines, Illinois
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - New Jersey Medical School, Newark, New Jersey
  - New York University School of Medicine, New York, New York
  - Columbia University/Presbyterian Medical Center, New York, New York
  - Harlem Hospital Center, New York, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Nashville VA Medical Center, Nashville, Tennessee
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Thomas Street Clinic, Houston, Texas
  - Audi L. Murphy VA Hospital, San Antonio, Texas
  - Seattle King County Health Department, Seattle, Washington
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Montreal Chest Institute McGill University, Montreal, Quebec

REFERENCES:
- [Background] Weiner M, Benator D, Burman W, Peloquin CA, Khan A, Vernon A, Jones B, Silva-Trigo C, Zhao Z, Hodge T; Tuberculosis Trials Consortium. Association between acquired rifamycin resistance and the pharmacokinetics of rifabutin and isoniazid among patients with HIV and tuberculosis. Clin Infect Dis. 2005 May 15;40(10):1481-91. doi: 10.1086/429321. Epub 2005 Apr 14. PMID 15844071
- See also: (Click here for more information about the Tuberculosis Trials Consortium(TBTC) — http://www.cdc.gov/nchstp/tb/tbtc/